CLINICAL TRIAL: NCT05993286
Title: Treatment of Misophonia: Comparison of Exposure and Sound Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kezban Burcu Avanoğlu, Consultant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16969557
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Misophonia
Keywords: Misophonia; sound therapy; exposure; psychoeducation; treatment
MeSH Terms: conditions — misophonia | interventions — Implosive Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of three groups: psychoeducation only (the active control group), exposure therapy with psychoeducation, and sound therapy with psychoeducation. All participants were assessed at baseline, and then at 3rd and 6th weeks. All of them received psychoeducation at study intake. A random one third received no further active treatment, one third received exposure, and one third received sound therapy.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psychoeducation (Other): This was an active control group and included information on the proposed mechanism of the development of misophonia, how symptoms are reinforced, and basic coping skills.
  Interventions: Other: Psychoeducation
- Exposure Therapy and Psychoeducation (Experimental): Exposure has been successfully used in the treatment of anxiety disorders, phobias, and obsessions. There are also case reports showing its effectiveness in the treatment of misophonia. The proposed procedure is to expose the misophonic person to the triggering sound in a controlled and gradual manner until habituation/desensitization to the trigger occurs. In the current research setting, each participant was asked to choose the two misophonic sounds that are most disturbing.
  Interventions: Behavioral: Exposure Therapy; Other: Psychoeducation
- Sound Therapy and Psychoeducation (Active Comparator): The music used in the current study was adapted from the protocol used by Jastreboff and Jastreboff (2013) for the treatment of misophonia. It includes noises such as white (noise with equal volume in all octaves) or pink noise (noise that decreases by 3 dB per octave towards high frequencies) or relaxing instrumental music
  Interventions: Other: Sound Therapy; Other: Psychoeducation

INTERVENTIONS:
Behavioral: Exposure Therapy — At Week 0, the homework was to expose oneself to these sounds for 20 minutes a day, three days a week for three weeks.
  At the Week 3 interview, the frequency and severity of the homework were adjusted based on the degree of improvement in the symptoms and the person's adherence to the instructions.
  Arms: Exposure Therapy and Psychoeducation
Other: Sound Therapy — Participants were asked to listen to specifically modulated music for twenty minutes a day, three days a week, for the first three weeks. At the Week 3 assessment, if the patient reported no or little benefit in their misophonia symptoms, the instruction was modified (intensified) to listening to the same music for forty minutes a day, three days a week.
  Arms: Sound Therapy and Psychoeducation
Other: Psychoeducation — A psychoeducation session, prepared by the research team was delivered by the investigator to each patient at the study intake.

SUMMARY:
The goal of this clinical trial is to compare the effects of possible treatments in misophonics. The main question it aims to answer is:

- Is exposure more effective on misophonic symptoms than sound therapy? Participants are randomly assinged to three groups of treatment;

1. Psychoeducation
2. Psychoeducation + Exposure
3. Psychoeducation + Sound Therapy

ELIGIBILITY:
Inclusion Criteria:

* People have Misophonia

Exclusion Criteria:

* Current psychosis
* Mental retardation or dementia
* those who had previously received exposure or sound therapy for misophonia symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
The mean change in Misophonia Total Score (MTS) | Week 0 and Week 6
  The difference between MTS Week 0 and MTS Week 6 was calculated, divided by MTS Week 0, and multiplied by 100, to elicit the percent change in MTS between Week 0 and Week 6.
The "improvement" | Week 3 and Week 6
  It was rated by the investigator (KBA) based on her clinical judgement (0=some worsening, 1=no improvement, 2=some improvement, 3=moderate improvement, 4=much improvement). If there was a moderate to much improvement at any point, the case was rated as "improved"; and "not improved" if the score was little worsening, no improvement, or some improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Cengiz Kılıç, Prof., Study Director — Hacettepe University
Locations (1):
- Hacettepe University Department of Psychiatry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swedo SE, Baguley DM, Denys D, Dixon LJ, Erfanian M, Fioretti A, Jastreboff PJ, Kumar S, Rosenthal MZ, Rouw R, Schiller D, Simner J, Storch EA, Taylor S, Werff KRV, Altimus CM, Raver SM. Consensus Definition of Misophonia: A Delphi Study. Front Neurosci. 2022 Mar 17;16:841816. doi: 10.3389/fnins.2022.841816. eCollection 2022. PMID 35368272
- [Background] Kilic C, Oz G, Avanoglu KB, Aksoy S. The prevalence and characteristics of misophonia in Ankara, Turkey: population-based study. BJPsych Open. 2021 Aug 6;7(5):e144. doi: 10.1192/bjo.2021.978. PMID 34353403
- [Result] Jager IJ, Vulink NCC, Bergfeld IO, van Loon AJJM, Denys DAJP. Cognitive behavioral therapy for misophonia: A randomized clinical trial. Depress Anxiety. 2020 Dec 18;38(7):708-18. doi: 10.1002/da.23127. Online ahead of print. PMID 33336858